CLINICAL TRIAL: NCT03009240
Title: A Phase I Study of Pevonedistat (TAK-924) and Decitabine Combination Therapy in High Risk Acute Myeloid Leukemia
Brief Title: Pevonedistat and Decitabine in Treating Patients With High Risk Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16270; NCI-2016-02044 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16270 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2016-12-30; First posted 2017-01-04 (Estimated); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Therapy-Related Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Injections; pevonedistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pevonedistat, decitabine) (Experimental): Patients receive pevonedistat IV over 1 hour on days 1, 3, and 5 and decitabine IV over 1 hour on days 1-5 and 8-12. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unexpected toxicity.
  Interventions: Drug: Decitabine; Other: Laboratory Biomarker Analysis; Drug: Pevonedistat; Other: Pharmacological Study

INTERVENTIONS:
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2''-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pevonedistat — Given IV
  Other Names: MLN4924; Nedd8-Activating Enzyme Inhibitor MLN4924
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of pevonedistat when given together with decitabine in treating patients with high risk acute myeloid leukemia. Pevonedistat and decitabine may stop the growth of cancer cells by blocking some of the enzymes need for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if the addition of pevonedistat to standard dose decitabine is safe and tolerable by the evaluation of toxicities including: type, frequency, severity, attribution, time course, reversibility and duration.

II. Determine the maximum tolerated dose (MTD)/recommended phase II dose (RP2D) of pevonedistat when given in combination with standard dose decitabine.

SECONDARY OBJECTIVES:

I. Obtain preliminary estimates of complete remission (CR) rate, overall response rate (ORR: CR+CRi [incomplete CR]), duration of response, and survival probabilities: overall survival (OS) and event-free survival (EFS) at 1-year and 2-years.

II. Demonstrate down-modulation of micro ribonucleic acid (miR)-155 and increased expression of miR-155 targets (SHIP1 and PU.1) in vivo.

III. Examine the impact of the combination on leukemia stem cells (LSCs); enriched blast cell subpopulations.

IV. Evaluate possible associations between changes in levels of miR-155, miR-155 gene targets (PU.1, SHIP1) and toxicity and/or clinical response.

OUTLINE: This is a dose-escalation study of pevonedistat.

Patients receive pevonedistat intravenously (IV) over 1 hour on days 1, 3, and 5 and decitabine IV over 1 hour on days 1-5 and 8-12. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unexpected toxicity.

After completion of study treatment, patients are follow up for 30 days, monthly for 1 year, and bi-monthly for another year.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute myeloid leukemia (AML) by World Health Organization (WHO) classification, meeting one of following criteria:

  * Age 60 or older, newly diagnosed, untreated, who are unwilling to undergo or not candidates for conventional induction chemotherapy with cytarabine/anthracyclines
  * Age 60 or older with relapsed or refractory disease
  * Younger adult patients with previously untreated high-risk disease (complex karyotype, inv[3] or t[3;3], t[6;9], monosomal karyotype, therapy-related and secondary disease) that are unwilling to undergo or not candidates for conventional induction chemotherapy with cytarabine/anthracyclines and/or allogeneic stem cell transplantation
  * Younger patients with refractory/relapsed AML who are otherwise not candidates for allogeneic stem cell transplantation
  * Patients with extramedullary disease who meet one of the above criteria may be included
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients with co-morbid medical illness, life expectancy attributed to this must be greater than 6 months
* The effects of pevonedistat and decitabine on the developing fetus is unknown; for this reason, women of child bearing potential and men must agree to use effective contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for 4 months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Female patients must be:

  * Postmenopausal for at least 1 year before the screening visit, OR
  * Surgically sterile, OR
  * If they are of childbearing potential

    * Agree to practice 1 highly effective method and one additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug (female and male condoms should not be used together), OR
  * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception)
* Male patients, even if surgically sterilized (i.e., status post-vasectomy) must:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 6 months after the last dose of study drug (female and male condoms should not be used together), or
  * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception)
* Creatinine < 1.5 X institutional upper limit of normal
* OR creatinine clearance >= 60 mL/min for patients with creatinine levels above 1.5 X institutional upper limit of normal
* Cardiac ejection fraction >= 50%
* Albumin > 2.7 g/dL
* Total bilirubin =< institutional upper limit of normal (ULN) (except in patients with Gilbert's syndrome; patients with Gilbert's syndrome may enroll if direct bilirubin is =< 1.5 x ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 ULN unless higher levels are related to leukemic infiltration
* Hemoglobin > 8 g/dL; patients may be transfused to receive this value; elevated indirect bilirubin due to post-transfusion hemolysis is allowed
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* The following patients are allowed:

  * Patients may have been treated for AML or antecedent hematologic disorder with myeloid growth factors, recombinant erythropoietin, thalidomide, lenalidomide, 5-azacitidine or decitabine
  * Any prior chemo therapy must have been completed >= 2 weeks prior to day 1 of study treatment and the participant must have recovered to eligibility levels from prior toxicity
  * There is no limit for prior chemo regimens
  * Patients may have received hematopoietic stem cell transplantation for AML or other diseases
  * Hydroxyurea is allowed prior to day 1 of study treatment for count control and during cycle 1; the use of hydroxyurea is not allowed beyond completion of cycle 1

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pevonedistat or decitabine
* Patients have received prior chemotherapy or radiation for AML < two weeks before study enrollment, or those who have not recovered from the adverse events due to agents administered
* Females who are both lactating and breastfeeding or who have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on day 1 before first dose of study drug
* Patients with additional (other than AML) active malignancies, other than curatively treated carcinoma in situ (CIS) of the cervix, or basal or squamous cell carcinoma of the skin; patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy and disease free from prior malignancies for > 2 years
* Life-threatening illness unrelated to cancer
* Known cardiopulmonary disease defined as one of the following:

  * Unstable angina
  * Uncontrolled high blood pressure (ie, systolic blood pressure > 180 mm Hg, diastolic blood pressure > 95 mm Hg)
  * Cardiomyopathy or history of ischemic heart disease
  * Arrhythmia (eg, history of polymorphic ventricular fibrillation or torsade de pointes); permanent atrial fibrillation (a fib) defined as a fib >= 6 months; persistent a fib defined as sustained a fib lasting > 7 days and/or requiring cardioversion in the 4 weeks before screening; however, patients with < grade 3 atrial fibrillation (a fib) for a period of at least 6 months may enroll; grade 3 a fib is symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation; patients with paroxysmal a fib are permitted to enroll
  * Implantable cardioverter defibrillator
  * Congestive heart failure (New York Heart Association [NYHA] class III or IV; or class II with a recent decompensation requiring hospitalization or referral to a heart failure clinic within 4 weeks before screening),
  * Myocardial infarction and/or revascularization (eg, coronary artery bypass graft, stent) within 6 months of first dose of study drug
  * Patients who had ischemic heart disease who have had ACS, MI, and/or revascularization greater than 6 months before screening and who are without cardiac symptoms may enroll
  * Moderate to severe aortic and/or mitral stenosis or other valvulopathy (ongoing)
  * Pulmonary hypertension
* Patients with uncontrolled coagulopathy or bleeding disorder
* Prolonged rate corrected QT (QTc) interval of > 500 msec, calculated according to institutional guidelines
* Left ventricular ejection fraction (LVEF) < 50% as assessed by echocardiogram or radionuclide angiography
* Known moderate to severe chronic obstructive pulmonary disease (COPD), interstitial lung disease, and pulmonary fibrosis
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of study procedures
* Treatment with any investigational products within 14 days before the first dose of any study drug
* Active uncontrolled infection or severe infectious disease, such as severe pneumonia, meningitis, septicemia, or methicillin resistant Staphylococcus aureus infection
* Major surgery within 14 days before the first dose of any study drug or a scheduled surgery during study period
* Known central nervous system (CNS) involvement
* Known human immunodeficiency virus (HIV) seropositive
* Known hepatitis B surface antigen seropositive or known or suspected active hepatitis C infection; Note: Patients who have isolated positive hepatitis B core antibody (ie, in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load; patients who have positive hepatitic C antibody may be included if they have an undetectable hepatitis C viral load
* Known hepatic cirrhosis or severe pre-existing hepatic impairment
* Systemic antineoplastic therapy or radiotherapy for other malignant conditions within 14 days before the first dose of any study drug, except for hydroxyurea
* White blood cell (WBC) > 50,000/mcL
* Treatment with clinically significant metabolic enzyme inducers within 14 days before the first dose of the study drug; clinically significant metabolic enzyme inducers are not permitted during this study (CYP3A4/5 inducers)
* Female patients who intend to donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s)
* Male patients who intend to donate sperm during the course of this study or 4 months after receiving their last dose of study drug(s)
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-08-21 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse effect assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03 | Up to 2 years
  Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.
Dose limiting toxicities (DLT) defined as any toxicities that are at least possibly related to pevonedistat that occur during cycle 1 assessed by NCI CTCAE version 4.03 | Up to 28 days
  Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.
Maximum tolerated dose (MTD) based on assessment of DLT | Up to 28 days
  Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.

SECONDARY OUTCOMES:
Complete remission (CR) rate assessed by International Working Group criteria | Up to 2 years
  Will be calculated as the percent of evaluable patients that have confirmed CR.
Overall response rate (ORR) (CR + incomplete CR [CRi]) assessed by International Working Group criteria | Up to 2 years
  Will be calculated as the percent of evaluable patients that have confirmed CR or CRi.
Overall survival (OS) | Time from start of study therapy until death, or last contact, whichever comes first, assessed up to 2 years
Event-free survival (EFS) | Time from start of study therapy until death, relapse/progression, receipt of anti-leukemia therapy, or last contact, whichever comes first, assessed up to 2 years
Duration of response | Time interval from the date of first documented response (CR or CRi) to documented disease relapse or death whichever occurs first, assessed up to 2 years

OTHER OUTCOMES:
miR-155 expression | Up to 2 years
miR-155 target gene (SHIP1 and PU.1) expression | Up to 2 years
NF-kappaB enrichment on miR-155 promoter | Up to 2 years
NF-kappaB activity | Up to 2 years
  Will be measured by gene reporter assays.
Nuclear NF-kappaB expression | Up to 2 years
  Will be measured by immunoblotting.
miR-155 promoter methylation | Up to 2 years
Leukemia stem cell (LSC) activity (LTC-IC frequency and activity in vitro and serial transplant experiments of LSC-enriched cell fractions) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Guido Marcucci, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States